CLINICAL TRIAL: NCT00830830
Title: A Double-Blind, Randomized Trial of Intra-Articular Injections of 20mg of Hyalgan for the Treatment of Knee Pain Due to Osteoarthritis (Three Injection Regimen for Efficacy and Duration - 20mg/2ml Dose) - Extension Study
Brief Title: TREAD-20 Extension - Treatment of Knee Pain Due to Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L_9385EXT
Record Dates: First submitted 2009-01-21; First posted 2009-01-28 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Hyaluronic Acid

INTERVENTIONS:
Drug: Hyalgan (sodium hyaluronate)

SUMMARY:
This extended study will evaluate the efficacy and safety of intra-articular injections of 20mg/2ml dose HYALGAN in patients with pain due to osteoarthritis (OA) of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Patients having given their written informed consent, prior to participating in the trial.
* Patients of either sex >= 40 years of age and of sufficient good health that they will be able to complete the 6-month follow-up.
* Patients with signs and symptoms of osteoarthritis of at least one knee:

  * Diagnosed according to ACR criteria.
  * Based upon a knee X-ray performed within 6 months prior to Screening, the radiograms must be classified as a Grade II or III for osteoarthritis of the knee according to the Kellgren & Lawrence grading system based upon a radiologist's written report or individual certified for reading knee radiograms. (Sharpening of the tibial spine is not considered to be an osteophyte).
* Patients with symptoms consistent with osteoarthritis of the knee for at least 6 months prior to Screening. These symptoms must include knee joint pain, and may include crepitus, swelling and/or effusion of the knee.
* At Screening, patients on any analgesic/anti-inflammatory medication should have a visual analogue scale (VAS) pain score after walking on a 50 ft flat surface of > 30 mm but < 90 mm using a 100 mm scale. If patients are not taking any analgesic/anti-inflammatory medication or have not taken any pain medication (prescription [Rx] or over-the-counter [OTC]) in the previous 3 days from Screening then they should have a VAS pain score after walking on a 50 ft flat surface of > 40 mm but < 90 mm. If bilateral knee pain is present, the investigator will select the more painful knee.
* At Screening and Baseline, if there is bilateral OA of the knee involvement, patients must have a VAS pain score for walking on a 50 ft flat surface of < 30 mm in the less painful contralateral knee at the Baseline assessment. A patient scoring an acceptable VAS pain score at Screening but failing to meet the inclusion and exclusion criteria at Baseline can not be randomized and enrolled.
* At Baseline, after all analgesic/anti-inflammatory medications have been discontinued for 2 weeks (withdrawal from acetaminophen rescue medication for at least 24 hours prior to Baseline assessment), patients should have a VAS pain score of > 40 mm but < 90 mm immediately after the 50-foot walk on a flat surface. Again, if bilateral knee pain is present, the investigator will select the more painful knee and the contralateral knee must have a VAS pain score of < 30 mm.
* Patients must have had knee pain in the signal knee on at least 50% of the days in the month preceding Screening.
* Patients who are able to complete efficacy measurement questionnaires and can understand and read English or Spanish (Spanish forms will be provided).
* Patients who can perform the 50-foot walk test without the support of crutches or other assistive devices, except for canes. If patient uses a cane routinely in daily activities, then they can use it for their assessments. However, this use must remain stable for all assessments.
* Minimum flexion of 90 degrees in both knees.
* Patients who are willing to discontinue all non-steroidal anti-inflammatory drugs (NSAIDs) or other analgesic medication taken for any condition, including their knee pain with the exception of acetaminophen, up to 1000 mg (2 tablets) four times a day (q.i.d.), as needed (p.r.n.) (maximum 8 tablets or 4 grams per day). These patients must be willing to use only acetaminophen as a rescue pain medication for the knee pain during the study period and refrain from even acetaminophen use 24 hours prior to any office visit. All other analgesic medications for any chronic condition must be stopped (see exceptions for acute treatment of transient flares of pain). Patients must also be willing to abstain from any intra-articular (i.a.) or peri-articular injections to the knee or surgery during the course of the trial, except for the assigned study product.
* Patients who, if they are currently taking low dose aspirin (325 mg/day or less), are willing to remain on a stable dose throughout the study and are willing to refrain from any aspirin dose 24 hours prior to any office visit.

Exclusion Criteria:

* Women of childbearing potential may not be entered if:

  * their pregnancy tests (urine test) are positive,
  * they are nursing,
  * they do not use an effective method of contraception until all follow-up procedures are complete. (Methods of contraception considered effective are an oral, injectable or implanted contraceptive agent, or an intra-uterine device with a failure rate of 1% per year, and abstinence).
* Patients participating in an experimental drug/device study or any clinical trial within the previous 30 days prior to Screening.
* Patients with a prior history of any malignancy with the exception of basal cell carcinoma of the skin treated more than 2 years prior to Screening, unless specific permission/waiver by the Sponsor is granted.
* Patients having significant bleeding diathesis.
* Patients that are currently under litigation for injuries related to the study knee or other injuries that might interfere with their completion of the study protocol.

Musculoskeletal Related

* Patients having any major injury (including sports) to the study knee in past 12 months.
* Patients having any surgery to the study joint within the previous 12 months prior to Screening, and surgery to the contralateral knee or other weight-bearing joint if it would interfere with the study assessments.
* Patients having significant surgery of lower limbs (hip, ankle, foot) that may interfere with knee assessments.
* Patients receiving any articular procedures, such as transplants, to the study knee.
* Patients having a ligament reconstruction to the study knee.
* Patients with inflammatory arthropathies such as rheumatoid arthritis, lupus, or psoriatic arthritis
* Patients with gout or calcium pyrophosphate (pseudogout) diseases that had flared within the previous 6 months prior to Screening.
* Patients receiving any intra-articular or local peri-articular corticosteroid injections to the study joint/knee within the previous 3 months prior to Screening.
* Patients receiving any intra-articular, intra-muscular or local peri-articular corticosteroid injections to any other joint (beside the study joint) or soft tissue area within the past 3 months.
* Patients receiving any oral corticosteroid within the previous month. Steroid inhalants are permitted if the patient has been on a stable regimen for the past month prior to Screening and remains on this regimen throughout the course of the trial.
* Patients receiving an intra-articular hyaluronan in the study joint within the previous 9 months prior to screening.
* Patients receiving an intra-articular hyaluronan in any joint within the previous 6 months prior to screening.
* Patients with a history of allergic reaction to an intra-articular injection or avian products.
* Patients taking unstable doses of glucosamine- or chondroitin sulfate-containing compounds, or patients taking stable dose for less than 4 months prior to Screening, or patients taking stable dose for at least 4 months prior to and unwilling to remain on these stable doses throughout the course of the trial.
* Patients on unstable doses of bisphosphonate or patients on stable doses for the past month prior to Screening, and are unwilling to remain on these stable doses throughout the course of the trial.
* Patients who cannot perform the 50-foot walk test without the support of crutches or other assistive devices, except for canes. If patient uses a cane routinely in daily activities, then they can use it for their clinical assessments. If the patient uses a cane for their Baseline assessment then they must use the cane for ALL subsequent assessments.
* Patients with X-ray findings of acute fractures, severe loss of bone density, avascular necrosis and/or severe bone or joint deformity.
* Patients with significant axial deviation of the knee.
* Patients with OA that is dominantly in the lateral compartment or any significant valgus deformity
* Patients with significant anterior knee pain due to diagnosed isolated patella-femoral syndrome or chondromalacia.
* Patients with symptomatic osteoarthritis of either hip, contralateral knee or spine that may interfere with functional assessment of the signal knee.
* Patients with clinically significant medio-lateral and/or anterior-posterior instability.
* Patients with osteonecrosis of either knee.
* Patients that are receiving or performing physical therapy regimen during the previous month from Screening, and/or will not or cannot maintain a stable physical therapy regimen throughout the course of the trial.
* Patients with Kellgren-Lawrence Grade IV OA (i.e., large osteophytes, marked narrowing, severe sclerosis, and definite deformity) and Grade I OA of the knee.
* Patients having any arthrogram of the signal joint within the past 3 months prior to Screening.
* Patients with a hemiparesis of the lower limbs
* Patients with active liver or renal disease based upon liver profile of SGOT > 2 x ULN (upper limit of normal), and/or conjugated bilirubin > 2 x ULN, and/or renal insufficiency (serum creatinine < 2.0 mg/dL, and/or any clinically significant laboratory value based on clinical history which the investigator feels may affect the evaluation of the patient.

Concomitant conditions, diseases, medications and/or clinical history

* Patients requiring chronic use of analgesia for pain (including pain in the other knee or any other joint) that may interfere with the evaluations of the test knee (such as possible use of rescue medication for these other conditions).
* Patients with known allergies to acetaminophen, lidocaine, hyaluronans, or avian products.
* Patients with a recurrent medical history of severe allergic or immune-mediated reactions.
* Patients with active infection of the skin near the potential injection site.
* Patients with any dermatological disease overlying the signal joint that would contraindicate multiple injections or aspirations.
* Patients taking any agent reported to have symptom relief for arthritis or be a disease/structure modifying drug (e.g. doxycycline, long-term tetracycline, s-adenosylmethionine [SAM], dimethyl sulfoxide [DMSO], dietary supplements or any herbal remedy taken for arthritic and joint conditions within the past month. Exceptions are products containing glucosamine/Chondroitin/ methylsulfonylmethane (MSM) if stable for 4 months prior to Screening and remain stable throughout study and fulfill the VAS pain entry criteria).
* Patients with peripheral neuropathy that would be severe enough to interfere with the evaluation of the patient.
* Patients with vascular insufficiency of lower limbs that is severe enough to interfere with the evaluation of the patient.
* Patients on concomitant therapy with anticoagulants (low dose aspirin, not exceeding 325 mg per day as an anti-thrombotic agent is permitted if stable for one month prior to Screening and remains stable throughout the study.
* Patients with any inter-current disease(s) or condition(s) that may interfere with the free use and evaluation of the affected knee for the 6 month course of the trial (cancer, other rheumatic diseases, gout, severe congenital defects, etc.).
* Patients with any inter-current chronic disease(s) or condition(s) that may predispose them to a high probability of interfering with the completion of the 6 month follow-up of the study such as peptic ulcer, liver disease, severe coronary disease, renal disease, cancer, pregnancy, alcoholism, drug abuse, mental state, or other clinically significant condition.
* Patients with excessive alcohol consumption or alcoholism that would be contraindicated with the use of acetaminophen.
* Patients with any known current addiction to pain medications.
* Patients that have, in the opinion of the clinical investigator, a clinically significant diagnostic test and/or abnormal laboratory test result(s) that may place the patient at a health risk, impact the study, or affect the patient's ability to complete the study.
* Patients unable to or with any psychiatric illness that would prevent them to legally comprehend the details and nature of the study.
* Patients who in the judgment of the clinician are likely to violate the protocol regulations or unlikely to complete the study for any reason.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-12; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Improvement in pain due to OA of the knee after 50-foot walk on a flat surface based upon 100 mm VAS score for up to 6 months after Baseline for the HYALGAN treated group compared to PB-Saline control

CONTACTS AND LOCATIONS:
Overall Officials: Tara Semanchik, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Inc, Bridgewater, New Jersey, United States

REFERENCES:
- See also: clinicaltrials.gov — http://clinicaltrials.gov/ct2/show/NCT00130468?term=L_9385&rank=1